CLINICAL TRIAL: NCT06807866
Title: Use of Duloxetine for Perioperative Pain Control After Total Hip Arthroplasty: Randomized Controlled Clinical Trial (RCT)
Brief Title: Duloxetine for Perioperative Pain in Hip Arthroplasty: A RCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20240579
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: THA
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duloxetine group (Experimental): Participants will be in this group for up to 2 hours.
  Interventions: Drug: Duloxetine
- Placebo group (Placebo Comparator): Participants will be in this group for up to 2 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Duloxetine — Participants will come in person and receive a one time 60 mg dose by mouth.
  Arms: Duloxetine group
Other: Placebo — Participants will come in person and receive a one time 60 mg placebo pill dose by mouth.
  Arms: Placebo group

SUMMARY:
The primary objective of this study is to compare total narcotic intake standardized via milligram morphine equivalents between duloxetine and placebo cohorts after a total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients undergoing primary total hip arthroplasty
* Ambulatory patient prior to fracture
* Subjects must be capable of providing informed consent
* English or Spanish speaking

Exclusion Criteria:

* Previous hemiarthroplasty or THA on ipsilateral hip
* History of Complex Regional Pain Syndrome in ipsilateral extremity
* History of demyelinating disorder or neurologic deficit that may contribute to altered pain tolerance or sensation
* Acute or chronic hip infection in ipsilateral extremity
* Pregnant or breastfeeding
* Open fracture
* Polytrauma
* Intravenous or drug users within 6 months of surgery
* Liver Failure via clinical diagnosis or international normalized ratio greater than 1.5 or partial thromboplastin time greater than 40
* Patients on selective serotonin reuptake inhibitor, serotonin norepinephrine reuptake inhibitor, monoamine oxidase inhibitor, and/or tricyclic anti-depressant
* Severe renal dysfunctions, such as glomerular filtration rate less than 30
* Moderate to severe depression as diagnosed by a clinician
* Taking cytochrome P450 1A2 inhibitors and cytochrome P450 1A6 inhibitors for the duration of 5 half-lives as these drugs are clinically eliminated within 5 half-lives
* History of uncontrolled narrow angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Total Milligram Morphine Equivalent (MME) | Up to 24 hours
  The primary outcome measure was milligram morphine equivalent units to measure pain intensity difference and total pain relief

SECONDARY OUTCOMES:
Change in Pain as measured by Visual Analog Scale (VAS) | Baseline, up to 24 hours, 3 months
  The VAS used for pain assessment consists of a line drawn in the form of a ruler, and numbers from 0 to 10 (with 0 as "no pain" and 10 as "unbearable pain") were asked to score.
Musculoskeletal function as measured by SMFA questionnaire | Up to 3 months
  The Short Musculoskeletal Function Assessment Questionnaire (SMFA) consists of 34 questions covering the assessment of the patients function and 12 questions related to how bothered patients are by their symptoms. All categories are scored together, totaling between 0-100 percent. The lower the score, the better the subject's function
Hospital Length of stay measured in hours | Up to 96 hours
  Hospital Length of stay measured in hours
Ambulation distance measured by meters | Up to 3 months
  Ambulation distance measured by meters

CONTACTS AND LOCATIONS:
Overall Officials: Victor Hernandez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No